CLINICAL TRIAL: NCT03686397
Title: A Phase III, Multicenter, Randomized, Double-Blind Clinical Trial to Assess the Efficacy and Safety of SVT-15652 Otic Solution Compared to Placebo for the Treatment of Fungal Otitis Externa (Otomycosis).
Brief Title: SVT-15652 Otic Solution for the Treatment of Otomycosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEAR-2
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-11

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SVT-15652 (Experimental): 1 vial twice daily
  Interventions: Drug: SVT-15652
- Placebo (Placebo Comparator): 1 vial twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SVT-15652 — 1 vial twice daily
  Other Names: SVT-15652 Otic Solution
  Arms: SVT-15652
Drug: Placebo — 1 vial twice daily
  Arms: Placebo

SUMMARY:
Multicenter, randomized, 2-arm parallel-group, double blind, placebo-controlled study in patients suffering from Otomycosis. This study will compare the efficacy and safety of SVT-15652 otic solution to that of Placebo, when administering one vial twice daily during 14 days.

ELIGIBILITY:
Main Inclusion Criteria:

* At least 18 years of age
* Clinical diagnosis of otomycosis in one or both ears, where topical treatment is indicated.
* Signs/symptoms of pruritus, otalgia and ear fullness.
* Debris or drainage clinically consistent with fungal infection.

Main Exclusion Criteria:

* Known bacterial otitis externa or malignant otitis externa.
* Tympanic perforation, tympanostomy tubes inserted and post mastoid surgery.
* Structural ear anomalies which may difficult the evaluation of the therapeutic response.
* Uncontrolled diabetes mellitus.
* Any infection requiring systemic antimicrobial or systemic antifungal therapy.
* Concomitant medicines that may interfere with the study evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator was an otolaryngologist.
Pre-assignment Details: A fungal culture was performed at baseline to know if subject had an ear infection due to Aspergillus or Candida spp.
  The main efficacy population of the study was the MITT population (evaluable patients): randomized subjects who had a positive baseline culture for Aspergillus spp and/or Candida spp.
  From the 194 subjects enrolled in the study, only 110 patients showed positive fungal culture for Aspergillus and/or Candida spp.
Groups:
- SVT-15652: Investigational treatment
- Placebo: Comparator
Period: Overall Study
Arm/Group | SVT-15652 | Placebo
Started (MITT Population) | 75 | 35
Completed | 70 | 27
Not Completed | 5 | 8
Not completed — Lack of Efficacy | 3 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — covid pandemic, bacterial ear culture | 2 | 0

BASELINE CHARACTERISTICS:
Population: MITT Population: Randomized patients who had positive baseline fungal culture for Aspergillus spp and/or Candida spp
Groups:
- Total: Total of all reporting groups
Arm/Group | SVT-15652 | Placebo | Total
Number analyzed (Participants) | 75 | 35 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.50) | 51.5 (15.78) | 52.4 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 15 | 50
  Male | 40 | 20 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 72 | 34 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Europe | 75 | 35 | 110

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Cure (Clinical and Mycological Cure)
Description: Percentage of subjects with therapeutic cure
Time Frame: Test of cure on day 24
Population: MITT Population: Randomized patients who had positive baseline fungal culture for Aspergillus spp and/or Candida spp
Measure: Count of Participants; unit: Participants
Arm/Group | SVT-15652 | Placebo
Number analyzed (Participants) | 75 | 35
Participants | 59 | 8

ADVERSE EVENTS:
Time Frame: Overall study period (about 4 weeks)
Description: If pre-existing signs and symptoms of otomycosis worsen during the study, this was considered a treatment failure instead of an adverse event.
  The adverse events were reviewed in the safety population which included subjects who received at least 1 dose of study medication (subjects could have positive or negative fungal culture at baseline because the results of baseline culture were not available until a few days after starting the study treatment).
Arm/Group | SVT-15652 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/127 | 1/64
Other Adverse Events (participants affected / at risk) | 0/127 | 3/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SVT-15652 (N=127) | Placebo (N=64)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SVT-15652 (N=127) | Placebo (N=64)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication shall be expressly authorized in written by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT03686397/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT03686397/SAP_001.pdf